CLINICAL TRIAL: NCT03007212
Title: Outcome of Transarterial Chemo-embolization (TACE) in Hepatocellular Carcinoma Patients With Partial Portal Vein Thrombosis
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Iman Fawzy Montasser, Associate professor of tropical medicine , Ain Shams university, Ain Shams University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Hepatocellular Carcinoma
Record Dates: First submitted 2016-12-24; First posted 2017-01-02 (Estimated); Last update posted 2017-01-02 (Estimated); Status verified 2016-12

CONDITIONS: Hepatocellular Carcinoma (HCC)
MeSH Terms: conditions — Carcinoma, Hepatocellular

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- HCC patients with Pranch portal vein thrombosis (Experimental): Thirty HCC patients (24 male, 6 females) Child A cirrhotics with branch PVT. Follow up was done at 1, 3, 6 and 12 months after first TACE. All patients underwent laboratory investigations including liver function tests to assess deterioration in liver functions, triphasic spiral CT to assess radiological response according to mRECIST criteria. Survival analysis was performed using Kaplan-Meier estimations.
  Interventions: Procedure: transarterial chemoembolization versus the standard treatment with sorafinib

INTERVENTIONS:
Procedure: transarterial chemoembolization versus the standard treatment with sorafinib — TACE procedures were performed by the interventional radiologist through femoral artery approach in all patients. Super-selective cannulation of the main feeders was performed using a microcatheter whenever possible. The c-TACE protocol consisted of intra-arterial infusion of cisplatin 50-100 mg mixed with lipiodol ,Just prior to injection, emulsion is prepared by intensive mixing of equal volumes of cytotoxic drug solution and iodized oil using the pumping method with two syringes and a three way stop cock. Injection is guided by fluoroscopy and results in dense accumulation of the emulsion within the tumor vascular bed. Injection of poor iodized oil up to a maximum volume of 10-20 cc is an option and is followed by embolization of feeding arteries by Gelfoam cubes .Endpoints of conventional TACE are complete filling of the tumor vascular bed with iodized oil and stop-flow in subsegmental and segmental feeding arteries..

SUMMARY:
Portal vein tumor invasion (PVT) is a common complication in HCC. the studyb Aimed to assess the outcomes after TACE in patients with branch PVT regarding Child classification, radiological response and 1 year survival.

DETAILED DESCRIPTION:
Thirty HCC patients (24 male, 6 females) Child A cirrhotics with branch PVT. Follow up was done at 1, 3, 6 and 12 months after first TACE. All patients underwent laboratory investigations including liver function tests to assess deterioration in liver functions, triphasic spiral CT to assess radiological response according to mRECIST criteria. Survival analysis was performed using Kaplan-Meier estimations.

ELIGIBILITY:
Inclusion Criteria:

* Patients with newly diagnosed HCC,
* Child class A and
* Portal vein branch tumoral thrombus (proved by imaging)
* written informed consent

Exclusion Criteria:

* patients with Child class B and C,
* main Portal vein thrombosis,
* previous management for HCC,
* Arterio-portal shunt
* refused to be enrolled

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2014-09; Primary Completion 2015-09 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
changes in Radiological Response in the (CT/ MRI) after the intervention | 1 year

IPD SHARING:
Plan to Share IPD: Undecided